CLINICAL TRIAL: NCT03084081
Title: A Randomized Controlled Trial Comparing Cure Rates of Cervical Intraepithelial Neoplasia Grade 2 and Higher (CIN2+) Treated With CO2-based Cryotherapy, CropPen, and Thermoablation (UH3)
Brief Title: An Innovative Treatment for Cervical Precancer (UH3)
Acronym: UH3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Basic Health International (Other); University of Southern California (Other); Instituto Salvadoreno del Seguro Social (Unknown); Hospital Universitario San Ignacio (Other); Medical College of Wisconsin (Other); Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-294; UH3CA189883 (NIH)
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Human Papilloma Virus (HPV); Cryotherapy; Thermoablation; Thermocoagulation; Low and Middle Income Countries (LMICs)
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CO2 standard therapy (Active Comparator): Double freeze treatment consists of three-minute freeze, five-minute thaw, three-minute freeze
  Interventions: Device: CO2 standard therapy
- CryoPen (Experimental): Single freeze treatment consists of one five-minute freeze
  Interventions: Device: CryoPen
- Thermocoagulator (Experimental): Thermoablation for 60-seconds at 100 degrees Celsius
  Interventions: Device: Thermocoagulator

INTERVENTIONS:
Device: CO2 standard therapy — Standard therapy using carbon dioxide for freezing of tissue
  Arms: CO2 standard therapy
Device: CryoPen — Provides a means of freezing tissue without the use of gases or liquids
  Arms: CryoPen
Device: Thermocoagulator — Thermoablation
  Arms: Thermocoagulator

SUMMARY:
The purpose of this academic-industrial partnership will compare the CryoPen® and thermoablator to traditional CO2-based cryotherapy for the treatment of cervical precancer in low and middle income countries (LMICs) and investigate whether the cure rates of cervical intraepithelial neoplasia 2 and more severe diagnoses (CIN2+) with these devices are non-inferior compared to that of conventional cryotherapy. The results of this study will affect other research areas by serving as a springboard to exploring treatment alternatives that are amenable to low-resource settings and thus will reach the most vulnerable populations.

DETAILED DESCRIPTION:
Cryotherapy is the current gold standard for treatment of precancerous cervical lesions in low resource settings. However, in recent years a number of issues-particularly the use of compressed gas, which requires storage and replenishment of large and potentially dangerous tanks-have emerged as clear limitations. Two technologies-the LMICs-adapted CryoPen®, manufactured and sold by CryoPen®, Inc. (TX, USA), and the thermoablator commercialized by WISAP Medical Technology (Germany) are treatment options for precancerous cervical lesions that run on electricity and avoid the difficulties associated with compressed gas. The LMIC-adapted CryoPen® (hereafter, CryoPen®) differs from previous cryotherapy methods in that it does not require an external source of gas (a tank), since the gas for cooling is built into the system. Thermoablation (also called thermocoagulation) has been used since the 1970s for treatment of cervical lesions. This is treatment with a probe heated to temperatures of 100 to 120ºC. It is also an effective, inexpensive method that does not require high-level healthcare providers.

The purpose of this study is to conduct a randomized non-inferiority clinical trial to compare the CryoPen® and WiSAP thermoablator to CO2-based cryotherapy for the treatment of CIN2 or more severe diagnoses ("CIN2+") but excluding microinvasive or invasive cervical cancer. The primary objective is to compare CIN2+ cure rates after treatment with the LMIC-adapted CryoPen®, the WISAP thermoablator, and CO2-based cryotherapy.

Women will be recruited from the Salvadorian Social Security Hospital (ISSS) in San Salvador, El Salvador, La Liga Contra el Cancer in Lima, Peru and Hospital Universitario San Ignacio in Bogota, Colombia. All are referral sites for women with abnormal cytology.

The investigators will approach approximately 1,602 women with CIN2+ during a 2.5 year enrollment phase (30 months). Assuming an approximately 80% participation rate, approximately 1,281 women will be enrolled- 1,152 (90%) will be eligible for cryotherapy (i.e. no contraindications) and 129 will be ineligible and undergo alternative treatments. The investigators estimate that approximately 20% will be lost to follow-up at the twelve-month visit, so that complete data will be available on a total of 922 women (57.55% of 1,602) treated with either CO2-based cryotherapy, LMIC-adapted CryoPen®, or thermoablation.

Eligible women with biopsy-confirmed CIN2+ will undergo HPV genotyping with next-generation sequencing. The specimen is taken prior to treatment to establish a baseline of which HPV types are present. If a different HPV type is present in the post-treatment specimen, this will be classified as a new rather than persistent infection. Testing will be conducted at the National Cancer Institute in Rockville, MD. Women will be randomly assigned to one of three study arms:

A. CO2-based cryotherapy (double freeze), B. CryoPen® (single freeze), or C. Thermoablation for 40 seconds at 100ºC.

At a pre-treatment visit, consented women will receive a pregnancy test as part of the eligibility criteria for enrollment in the study. Pre-vaginal cultures will be collected to be analyzed for bacterial vaginosis, yeast, gonorrhea and chlamydia. The same cultures will be collected at a 6-week follow-up visit. Consented women will be enrolled and undergo a pelvic exam and visual inspection of the cervix following placement of diluted acetic acid on the cervix. Images of the cervix will be taken with a mobile ODT device will be taken before and after treatment. Women deemed ineligible for cryotherapy will undergo LEEP immediately. In the case of suspected cancer, women will be appropriately referred.

Six weeks post-treatment, women who return for a visit for evaluation of treatment side effects; these women will complete a questionnaire to assess the presence of pain or cramps, bleeding, stenosis, watery discharge, malodorous discharge and be evaluated for evidence of cervicitis. In addition, vaginal cultures will be collected and analyzed for bacterial vaginosis, yeast, gonorrhea, and chlamydia.

One year post-treatment, women will return for a follow-up visit to determine residual disease, which is the primary endpoint. Residual disease will be determined by colposcopy and four-quadrant biopsies. In addition, VIA, cytology, and high-risk HPV DNA testing with careHPV will be performed. Genotyping and next-generation sequencing will be repeated to differentiate between persistent and new infections. The goal is to evaluate sensitivity of VIA, cytology, and HPV testing post-treatment. Women diagnosed with recurrent/untreated CIN2+ on biopsy will be asked to return to undergo LEEP. Women with suspected cancer on biopsy will be referred to the local cancer hospital for standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and older
* Biopsy results of CIN2, CIN2-3, CIN3, or high-grade CIN not otherwise specified
* Willing and able to provide informed consent
* Willing and able to provide permanent or reliable address

Exclusion Criteria:

* Pregnant or plans to become pregnant during study
* History of total hysterectomy (verified by medical record or pelvic evaluation)
* Previous surgery destructive to the cervix within the last 5 years
* Patient not eligible for cryotherapy (lesion >75% of cervix, lesion extends into canal or there is suspicion for invasive cancer)
* Cervix shape disfigured or hard to reach

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1132 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Cremer, MD, Principal Investigator — The Cleveland Clinic
Locations (3):
- Shanxi Academy of Medical Sciences Shanxi Bethune Hospital, Taiyuan, China
- Hospital Universitario San Ignacio, Bogotá, Colombia
- Instituto Salvadoreno del Seguro Social (ISSS), San Salvador, El Salvador

IPD SHARING:
Plan to Share IPD: No
IDP data will not be shared at the completion of the study.

REFERENCES:
- [Derived] Soler M, Alfaro K, Masch RJ, Conzuelo Rodriguez G, Qu X, Wu S, Sun J, Hernandez Jovel DM, Bonilla J, Puentes LO, Murillo R, Alonzo TA, Felix JC, Castle P, Cremer M. Safety and Acceptability of Three Ablation Treatments for High-Grade Cervical Precancer: Early Data From a Randomized Noninferiority Clinical Trial. JCO Glob Oncol. 2022 Dec;8:e2200112. doi: 10.1200/GO.22.00112. PMID 36525620

RESULTS

PARTICIPANT FLOW:
Groups:
- Thermocoagulator: Thermal ablation for 40-seconds at 100 degrees Celsius and reapplied at 20 second applications to cover the entire transformation zone.
  Thermocoagulator: Thermoablation
Period: Overall Study
Arm/Group | CO2 Standard Therapy | CryoPen | Thermocoagulator
Started | 377 | 377 | 378
Completed | 332 | 332 | 344
Not Completed | 45 | 45 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CO2 Standard Therapy | CryoPen | Thermocoagulator | Total
Number analyzed (Participants) | 377 | 377 | 378 | 1132
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean age in years | 36.3 (9.6) | 36.9 (9.0) | 35.9 (8.9) | 36.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 377 | 377 | 378 | 1132
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 256 | 256 | 257 | 769
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 121 | 121 | 121 | 363
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Colombia | 31 | 31 | 31 | 93
  El Salvador | 90 | 90 | 90 | 270
  China | 256 | 256 | 257 | 769

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Residual CIN2+
Description: Diagnosis of recurrent and or untreated cervical intraepithelial neoplasia grade 2 or higher with cervical cancer diagnosis
Time Frame: 12-months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | CO2 Standard Therapy | CryoPen | Thermocoagulator
Number analyzed (Participants) | 377 | 377 | 378
Participants | 18 | 29 | 25

2. Secondary Outcome: Self-reported Pain
Description: Patient pain scores using the Wong-Baker FACES Pain Rating Scale from 0-10 where 0 represents the best outcome (no pain) and 10 represents the worst outcome (worst pain). The underlying construct is pain experienced by the participant.
Time Frame: Pain during treatment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | CO2 Standard Therapy | CryoPen | Thermocoagulator
Number analyzed (Participants) | 377 | 377 | 378
units on a scale | 2 [0 to 4] | 2 [0 to 4] | 4 [2 to 6]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | CO2 Standard Therapy | CryoPen | Thermocoagulator
All-Cause Mortality (participants affected / at risk) | 0/377 | 0/377 | 0/378
Serious Adverse Events (participants affected / at risk) | 1/377 | 0/377 | 0/378
Other Adverse Events (participants affected / at risk) | 167/377 | 143/377 | 64/378
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CO2 Standard Therapy (N=377) | CryoPen (N=377) | Thermocoagulator (N=378)
Hospitalization (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CO2 Standard Therapy (N=377) | CryoPen (N=377) | Thermocoagulator (N=378)
Vasovagal response (Nervous system disorders) | 138 (138) | 121 (121) | 24 (24)
Infection (Infections and infestations) | 29 (29) | 22 (22) | 40 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03084081/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT03084081/ICF_001.pdf